CLINICAL TRIAL: NCT01825811
Title: A Single-blind, Randomized, Parallel-group, Multi-center Phase 2 Study to Determine the Efficacy and Safety of TissueGene-C Mixed With Fibrin-glue in Patients With Degenerative Arthritis
Brief Title: Efficacy and Safety Study of TissueGene-C Mixed With Fibrin-glue for the Patients With Degenerative Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS-TGC(S)-01-2
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Degenerative Arthritis
Keywords: Cell mediated gene therapy; Osteoarthritis; Fibrin-glue; Degenerative Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TissueGene-C (Low dose) (Experimental): TissueGene-C (1.0 x 10^6 cells per cm^2 of the cartilage defect) combined with fibrin-glue
  Interventions: Biological: TissueGene-C (Low dose)
- Experimental: TissueGene-C (High dose) (Experimental): TissueGene-C (3.0 x 10^6 cells per cm^2 of the cartilage defect) combined with fibrin-glue
  Interventions: Biological: TissueGene-C (High dose)

INTERVENTIONS:
Biological: TissueGene-C (Low dose) — TissueGene-C at 1.0 x 10^6 cells mixed with fibrin-glue
  Arms: TissueGene-C (Low dose)
Biological: TissueGene-C (High dose) — TissueGene-C at 3.0 x 10^6 cells mixed with fibrin-glue
  Arms: Experimental: TissueGene-C (High dose)

SUMMARY:
The purpose of this study is to determine whether TissueGene-C, allogeneic human chondrocytes expressing Transforming Growth Factor(TGF)-b1, mixed with fibrin-glue is effective and safe in patients with degenerative arthritis.

DETAILED DESCRIPTION:
TissueGene-C is a biological new drug which consists of non-transduced chondrocytes and transduced chondrocytes that express TGF-b1 to regenerate the damaged cartilage.

During the clinical trial Phase 2, the investigators compare low dose or high dose TissueGene-C in 12 - months trial with 18 outpatients who have degenerative arthritis. The patients are randomized to two dose levels of TissueGene-C by 1:1 ratio, and they are monitored and recorded for alleviating symptoms, sports activities, function of the knee, and the presence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 years or more
2. Diagnosed with degenerative arthritis of the knee
3. With an IKDC score of 60 or lower at the screening visit
4. With a BMI of higher than18.5 and lower than 30
5. With an International Cartilage Repair Society(ICRS) Grade IV cartilage damage in the major lesions, as confirmed through an MRI scan
6. With major lesions concentrated in one section of the knee, and with the major lesions considered the main cause of the clinical symptoms
7. With major lesions defect size 2 cm2 ~ 10cm2
8. With no alleviation of the symptoms even after at least three months of non-surgical treatment
9. Healthy, with no major findings from the physical examination, hematology, serum chemistry, and urine tests, and no significant medical history
10. Agreed to use an effective contraceptive method during the study period
11. Voluntarily agreed to participate in this study, and signed the informed consent form

Exclusion Criteria:

1. Showed clinically significant hematology, serum chemistry, and urine test results at the screening visit
2. Mechanical axis (HKA) is greater than 5°
3. Patients receiving injections to the treated knee within 2 months prior to study entry
4. Patients who are pregnant or currently breast-feeding children
5. With another joint disease (e.g., inflammatory arthritis, infectious arthritis)
6. With an infectious disease, including HIV or hepatitis
7. With any of the following clinically significant diseases:

   * heart disease [e.g., myocardial infarction, arrhythmia, other serious heart diseases,
   * kidney disease (e.g., chronic renal failure, glomerulonephritis)
   * liver disease (e.g., liver cirrhosis, fatty liver, acute or chronic liver disease)
   * endocrine disease (e.g., hyperthyroidism, hypothyroidism, thyroiditis, diabetes insipidus, Cushing's disease)
   * insulin-dependent diabetes mellitus
   * medical history of past or current malignant tumor
   * In particular, the tumors that TissueGene-C may aggravate can be screened using the following tests:

     * Leukemia (White Blood Cell level in the hematology)
     * Osteochondroma, Chondromas, Chondroblastoma, Chondromyxoid fibroma, Chondrosarcoma(Alkaline phosphatase level in the hematology)
8. Participated in another clinical trial (using the investigational drug or a medical device) within 30 days before enrollment in this study
9. Considered inappropriate by the investigator for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in IKDC Subjective Knee Evaluation | Week 0 and 48
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)

SECONDARY OUTCOMES:
Changes in WOMAC scores | Week 0, 24 and 48
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)
Changes in KOOS scores | Week 0, 24 and 48
  Symptoms, pain and functionality of the knee joint will be evaluated via the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Changes in 100 mm-VAS | Week 0, 24 and 48
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)
Comparative Evaluation of Knee Magnetic Resonance Images (MRIs) | Week 0, 24 and 48
  Comparison of pre-procedure MRI scans to those obtained at pre-dosing and at months 6 and 12 by an independent radiographic reviewer
Changes in ICRS Cartilage Repair Assessment | week 0 and 48
Changes in IKDC Subjective Knee Evaluation | Week 0 and 24
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)
Changes in KOOS QOL Sub-scale scores | Week 0, 24 and 48
Proportion of Patients Use of Rescue Medication | Week 12, 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Myung Chul Lee, MD, PhD, Principal Investigator — Seoul National University Hospital; Chul Won Ha, MD, PhD, Principal Investigator — Samsung Medical Center; Seong Il Bin, MD, PhD, Principal Investigator — Asan Medical Center; Myung Gu Kim, MD, PhD, Principal Investigator — Inha University Hospital; Jae Doo Yoo, MD, PhD, Principal Investigator — Ewha Womans University Mokdong Hospital; Hee Su Kyung, MD, PhD, Principal Investigator — Kyungpook National University Hospital
Locations (6):
- South Korea (6):
  - Kyungpook National University Hospital, Daegu
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul